CLINICAL TRIAL: NCT02985307
Title: Efficacy of Mobile Telehealth Short Message Service (SMS) as a Facilitator for Weight Management: A Randomised Controlled Trial
Brief Title: Impact of Mobile Phone Texting Service to Support Weight Loss
Acronym: SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Collaborators: Queen Margaret University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16/SS/0200
Record Dates: First submitted 2016-11-29; First posted 2016-12-07 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2019-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Message Text Service (Experimental): Participants receive short messages daily via their mobile phone
  Interventions: Behavioral: Short Message Text Service
- Standard Weight Management Group (Active Comparator): Participants attend standard group weight management sessions
  Interventions: Behavioral: Standard Weight Management Group

INTERVENTIONS:
Behavioral: Short Message Text Service — A service designed by professionals inside the National Health Service (NHS) to provide support and advice for participants to manage weight loss. It combines the expertise of the healthcare team and the convenience of the participant's own mobile phone to give prompts and advice to act on. It makes use of the familiar and convenient mobile phone text service 'SMS' to communicate directly with participants.
  Arms: Short Message Text Service
Behavioral: Standard Weight Management Group — A standard Lothian NHS group programme facilitated by a Dietitian
  Arms: Standard Weight Management Group

SUMMARY:
This study evaluates the efficacy of a mobile telehealth short message service as a facilitator for weight management. Half of the participants will receive a standard care weight management group intervention, while the other half will receive daily text messages via their mobile phone to help facilitate weight loss. It is hypothesized that the intervention group receiving text messages will be as successful as the control group at achieving weight loss over a 3-month period.

DETAILED DESCRIPTION:
Obesity, a chronic progressive disease, has become a major public health concern due to its increasing prevalence and association with many adverse health conditions including type 2 diabetes, many cancers and heart disease. The number of individuals requiring weight management intervention is increasing necessitating the need to explore other initiatives.

Developments in health technology are growing in popularity and there is increasing evidence that this type of intervention for obesity can significantly improve clinical outcomes. Mobile phones are a popular means of communication that provide a convenient, inexpensive means to deliver a health technology intervention.Short message service (SMS) by mobile phone has the potential to serve as an intervention medium to promote weight loss that is accessible and easy to use.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 35kg/m requiring to lose weight for an operation or having a co-morbidity including diabetes, osteoarthritis, high cholesterol, asthma, heart disease, high blood pressure or sleep apnoea or with a body mass >40kg/m with no co-morbidities.
* Own a mobile phone
* Have the ability to use short message service
* Have access to weighing scales
* Mentally capable of informed consent
* Have the ability to read and speak English

Exclusion Criteria:

* Uncontrolled Hypothyroidism
* Poorly controlled psychiatric illness
* Current alcohol or drug abuse
* Learning disability
* Do not own a mobile phone
* Do not have access to weighing scales
* Does not have the ability to read or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 3 months
  weight recorded in Kg on a Seca 635 medical digital load cell balance

SECONDARY OUTCOMES:
Behavioural changes necessary for weight loss | 3 months
  Self reported dietary and physical activity changes using 7-day food and exercise diaries
Body fat changes | 3 months
  Measured using a medically approved and validated scale: Tanita SC-240MA body composition analyser
Body Mass index | 3 months
  calculated using the formula weight in kg divided by height squared in metres
Height | 3months
  Height measured using Seca portable stadiometer with a sliding head plate

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McBean, PhD, Study Director — Queen Margaret University
Locations (2):
- United Kingdom (2):
  - Elizabeth McAnally, Edinburgh, West Lothian
  - NHS Lothian, Edinburgh, West Lothian

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for all primary and secondary outcome measures will be made available within 6months of study completion

REFERENCES:
- [Result] Patrick K, Raab F, Adams MA, Dillon L, Zabinski M, Rock CL, Griswold WG, Norman GJ. A text message-based intervention for weight loss: randomized controlled trial. J Med Internet Res. 2009 Jan 13;11(1):e1. doi: 10.2196/jmir.1100. PMID 19141433
- See also: World Health Organisation — http://www.comminit.com/global/content/mhealth-new-horizons-health-through-mobile-technologies